CLINICAL TRIAL: NCT05704998
Title: INVESTIGATION AND COMPARISON OF THE EFFECTS OF POSTURE EXERCISES ON DYSFUNCTION, POSTURE AND BALANCE IN INDIVIDUALS WITH POSTERIOR EDENTULOUS AND FULL-TOOTHED TEMPOROMANDIBULAR DISORDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Rübeysa Türedi, Physiotherapist, Dokuz Eylul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEU.HSI.MSc-2019970200
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Temporomandibular Disorder
Keywords: temporomandibular joint; physiotherapy; posture exercises; posterior tooth loss
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A total of 26 patients with temporomandibular disorder, aged between 18-70 years, 13 of whom were in the Posterior Edentulous Group (PDG) and 13 were in the Fully Toothed Group (TDG), received same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior Edentulous Group (Experimental): Posture exercises, manual therapy and kinesio taping were applied twice a week for six weeks.
  Interventions: Other: Physiotherapy
- Fully Toothed Group (Experimental): Posture exercises, manual therapy and kinesio taping were applied twice a week for six weeks.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Posture exercises, myofascial release techniques, sternocleidomastoideus and upper trapezius kinesio taping, trigger point ischemic compression, suboccipital release technique, cervical traction, deep neck flexors endurance exercises, massage
  Other Names: Manuel therapy; Kinesio taping

SUMMARY:
The aim of this study is to investigate the relationship between neck posture and balance in patients with posterior edentulous and full-toothed temporomandibular disorder and to compare the effectiveness of the physiotherapy program to be applied.

DETAILED DESCRIPTION:
The study was planned as a quasi-experimental controlled study. A total of 26 patients with temporomandibular disorder, aged between 18-70 years, 13 of whom were in the Posterior Edentulous Group (PDG) and 13 were in the Fully Toothed Group (TDG), were included. Posture exercises and manual therapy were applied to both groups twice a week for six weeks. Mandibular range of motion, pain, muscle strength, deep neck flexor endurance, flexibility, shortness, range of motion (ROM), pressure pain threshold (BAE), psychological state, posture and balance were evaluated before and after exercise.

The results of the study showed that six weeks of postural exercises and manual therapy provided significant improvement in all values (p<0.05). A significant difference was found in pain, muscle strength, ROM, BAE and balance in PDG compared to TDG (p<0.05).

The results of the study showed that symptoms can be improved by giving posture exercises in patients with tempromandibular disorder. It was concluded that the improvement in PDG was higher than in TDG.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Myofascial Temporomandibular Disorder according to The Research Diagnostic Criteria for Temporomandibular Disorders
* Complaining of head or neck pain
* Having temporomandibular joint pain for at least 3 months
* Not having used an intraoral plaque before
* Able to follow the treatment protocol regularly
* Ability and willingness to communicate verbally

Exclusion Criteria:

* Being positive for COVID-19
* Sports injuries
* Presence of trauma
* Whiplash
* Degenerative changes
* Signs or symptoms of disc displacement, osteoarthrosis or osteoarthritis of temporomandibular joint
* Post-operative conditions involving the cervical or temporomandibular region
* Burn involving the cervical region and the temporomandibular region
* Patients using analgesics or muscle relaxants up to 8 hours before the physical therapy procedure
* Those with hypermobility in cervical movements
* Those who have received physiotherapy or other treatment from the head / neck area in the last 12 months
* Acute infections or any systemic disorder
* Osteoporosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Mandibular Range of Motion | Baseline and week 6
  Maximal mouth opening, protrusion and both lateral excursions was recorded in millimeters.
  Change = ( Week 6 Score - Baseline Score) Comparison = (Posterior Edentulous Group Change Score - Fully Toothed Group Change Score)
Posture | Baseline and week 6
  Posture evaluated with New York Posture Rating Chart. Possible scores range from 13 (bad posture) to 65 (very good posture) Change = ( Week 6 Score - Baseline Score) Comparison = (Posterior Edentulous Group Change Score - Fully Toothed Group Change Score)
Balance | Baseline and week 6
  Balance evaluated with TETRAX® Interactive Balance System. Possible scores range from 0 (minimum fall risk) to 100 (high fall risk).
  Change = ( Week 6 Score - Baseline Score) Comparison = (Posterior Edentulous Group Change Score - Fully Toothed Group Change Score)

SECONDARY OUTCOMES:
Pain Score with Numeric Pain Rating Scale (NPRS) | Baseline and week 6
  NPRS is a validated, self-reported instrument assessing average pain intensity. Possible scores range from 0 (no pain) to 10 (worst possible pain).
  Change = ( Week 6 Score - Baseline Score) Comparison = (Posterior Edentulous Group Change Score - Fully Toothed Group Change Score)
Active Cervical Range of Motion | Baseline and week 6
  Measured by a phone app named Clinometer. Change = ( Week 6 Score - Baseline Score) Comparison = (Posterior Edentulous Group Change Score - Fully Toothed Group Change Score)
Beck Depression Inventory | Baseline and week 6
  Beck Depression Inventory, which is a validated, self-reported scale, consists of 21 questions. According to the total result, 0-9 points indicates minimal depression, 10-16 points mild depression, 17-29 moderate depression, 30-63 severe depression.
  Change = ( Week 6 Score - Baseline Score) Comparison = (Posterior Edentulous Group Change Score - Fully Toothed Group Change Score)

CONTACTS AND LOCATIONS:
Overall Officials: Selnur NARİN ARAL, Assoc. Dr., Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided